CLINICAL TRIAL: NCT06388057
Title: Intraoperative Ultrasound of Small Bowel in the Study of the Characteristics of the Surgical Resection Margin in Crohn's Disease
Brief Title: Intraoperative Ultrasound in Crohn's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5836
Record Dates: First submitted 2023-11-06; First posted 2024-04-29 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2023-11

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Patients with Crohn's disease with an indication for surgery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Crohn's disease with indication for surgery (Experimental)
  Interventions: Diagnostic Test: Intraoperative Small Bowel Ultrasonography

INTERVENTIONS:
Diagnostic Test: Intraoperative Small Bowel Ultrasonography — An intraoperative ultrasound study will be performed on the intestinal segment identified as the resection site

SUMMARY:
To study the role of intraoperative ultrasound of small bowel as a possible tool that can reduce the rate of histologically involved resection margins from Crohn's Disease.

DETAILED DESCRIPTION:
Patients with indication for resective surgery for Crohn's Disease will be enrolled and undergo to the planned surgery.

During surgery the site where to conduct the bowel resection will be decided according to the current indications in the literature and according to good clinical practice (absence of macroscopical signs of disease).

Before conducting the surgical resection, will be performed intraoperative ultrasonography of the small bowel at the intestinal segment chosen as the site of the resection.

Ultrasound features will be evaluated to determine whether or not there are any ultrasonographic signs ascribable to Crohn's Disease.

Once the above ultrasound has been completed (estimated time approximately 5-10 minutes), the predetermined resection will be conduct and the surgical piece will be sent for final histological examination as usual.

The outcome of intraoperative ultrasound will be schematized as positive or negative based on the presence or absence of specific ultrasound signs of intestinal inflammation attributable to Crohn's Disease.

The data will be collected and subsequently analyzed in order to compare the ultrasound findings acquired on the resection margins with the outcome of the histological examination conducted on the same site.

Patients will then enter a regular gastroenterological/surgical follow-up and undergo colonoscopy at 12 months after surgery as usual.

Data on clinical, surgical or endoscopic recurrence in the follow-up period will be collected and analyzed to compare the recurrence rate in the group of patients with intraoperative ultrasonographic features with the group without intraoperative ultrasonographic features on the resection margin.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 years or older.
* Confirmed diagnosis of Crohn's disease
* Indication for intestinal resection surgery for Crohn's Disease (first surgery or surgery for postoperative recurrence).

Exclusion Criteria:

* Patients who did not express their consent to participate in the study by signing the appropriate informed consent
* Patients younger than 12 years of age
* Patients with an indication for non-resective surgery for Crohn's Disease (e.g., ileostomy closure).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Specificity and sensibility of intraoperative ultrasound of small bowel in identifying resection margins histologically involved by Crohn's disease | 10 minutes
  To compare the number of ultrasound-positive resection margins with the number of histologically positive resection margins. This comparison will be conducted using basic statistics to determine the specificity and sensitivity of intraoperative ultrasound of the small bowel in identifying resection margins histologically involved by Crohn's disease.